CLINICAL TRIAL: NCT06155318
Title: 68Ga-DOTATOC PET for the Evaluation of Gastroenteropancreatic Neuroendocrine Tumours
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: PET-NET Prospective
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 68Ga-DOTATOC PET as a part of their clinical diagnostic work-up will be included — Patients meeting the inclusion criteria will undergo 68Ga-DOTATOC PET(PET/MRI or PET/CT) as part of their routine work-up, according to the referral clinicians' indication.PET/MRI will be performed on a 3.0T time of flight PET/MRI. Simultaneous PET/MRI will start approximately 60 minutes after the injection of 68Ga-DOTATOC.

SUMMARY:
Gastroenteropancreatic neuroendocrine tumours (GEP-NETs) are a heterogeneous group of neoplasms that arise from the endocrine cells of the gastroenteropancreatic tract.

The diagnostic work-up of these tumours include Computed Tomography (CT), Endoscopic Ultrasound (EUS), Magnetic Resonance Imaging (MRI).

The majority of these tumours express somatostatin receptors on their surface. For this reason, in addition to traditional imaging exams, diagnostic work-up of GEP-NETs should include a Positron Emission Tomography/CT with 68Ga labeled somatostatin analogues targeting somatostatin receptors with high sensitivity and specificity. 68Ga-DOTATOC PET/CT scan is a corner stone to assess GEP- NET patients at different stage of disease and it is the standard functional imaging modality to study well-differentiated Pan-NETs, as reported in the being also included in the guidelines of the European Association of Nuclear Medicine (EANM). Moreover, quantitative parameters extracted from 68Ga- DOTA-peptides PET imaging have demonstrated their prognostic utility as markers for progression-free survival and disease specific mortality in patients affected by NET.

Additionally, 18F-FDG PET can be used for evaluating the possible presence ofa high-grade component within the tumour itself. The accurate morphofunctional characterization is of utmost importance in the field of GEP-NET.

the advent of new hybrid scanners, namely PET/MRI, opens the way to an innovative diagnostic work- up that can be applied to GEP-NETs. In fact, MRI plays a role as morphological imaging modalities for a better characterization of soft-tissue and liver parenchyma compared to CT; moreover, the low radiation exposure related to MRI, makes this imaging modality more suitable for patients requiring several imaging during follow-up.

Patients requiring 68Ga-DOTA peptides (68Ga-DOTATOC) PET scan and eventually MRI scan, can be studied in a single session examination, by using 68Ga-DOTATOC PET/MRI.

Considering the rarity of GEP_NETs, it is quite difficult to collect a sufficient number of patients in order to investigate the accuracy, predictive and prognostic value of the currently available imaging technique in this scenario. Based on these considerations, the possibility to analyze PET images deriving from both PET/CT and PET/MRI scans of patients affected by GEP-NET is of fundamental relevance in order to provide answers to the currently unmet clinical needs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either histological diagnosis of GEP-NET at radiologic imaging and referred to 68Ga-DOTATOC PET;
* Age > 18 years old;
* Willing to provide a signed informed consent.

Exclusion Criteria:

* Controindications to MR study (i.e. Pacemaker);
* Age< 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Main selection criteria: patients with GEP-NET referred for 68Ga-DOTATOC PET.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2029-05-05 (Estimated); Study Completion 2029-05-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy | 10 years
  68GaDOTATOC PET in the identification of the site/s of disease in patients affected by neuroendocrine tumours, both in the staging and restaging phases.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No